CLINICAL TRIAL: NCT06435832
Title: Evaluation of the Effects of Tranexamic Acid and Chlorhexidine Gel on Alveolar Osteitis Incidence
Brief Title: Evaluations of the Effects of Tranexamic Acid and Chlorhexidine Gel on Alveolar Osteitis Incidence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Zeynep Gumrukcu, Associate Professor, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RTEUni
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Alveolar Osteitis
Keywords: Alveolar Osteitis
MeSH Terms: conditions — Dry Socket | interventions — Gelatin Sponge, Absorbable; Chlorhexidine; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- just absorbable gelatin (Active Comparator): After tooth extraction, only saline irrigation was applied and a absorbable gelatin sponge was placed in the socket.
  Interventions: Drug: Absorbable Gelatin
- absorbable gelatin with Chlorhexidine gel (Active Comparator): After tooth extraction, after irrigation with saline, 2% chlorhexidine gel was absorbed into gelatin sponges and placed into the socket.
  Interventions: Drug: Chlorhexidine
- absorbable gelatin with tranexamic acid (Active Comparator): Tranexamic acid 50mg/ml for injection after saline irrigation after tooth extraction solution into gelatin sponges was applied to the socket after it was cured.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Absorbable Gelatin — After tooth extraction, only saline irrigation was applied and a absorbable gelatin sponge was placed in the socket.
  Arms: just absorbable gelatin
Drug: Chlorhexidine — After tooth extraction, after irrigation with saline, 2% chlorhexidine gel was absorbed into gelatin sponges and placed into the socket.
  Arms: absorbable gelatin with Chlorhexidine gel
Drug: Tranexamic acid — Tranexamic acid 50mg/ml for injection after saline irrigation after tooth extraction solution into gelatin sponges was applied to the socket after it was cured.
  Arms: absorbable gelatin with tranexamic acid

SUMMARY:
This intervention is the treatment of alveolar osteitis (alveolitis) with different effects, which occurs due to the formation of clot after extraction, which is one of the most common intervals after tooth extraction.98 healthy patients with molar and premolar teeth with indication for extraction were taken to the Recep Tayyip Erdoğan University Faculty of Dentistry, Department of Oral and Maxillofacial Diseases and Surgery clinic between May 2024 and June 2024 (age: 38 sessions: 19). -62) 113 teeth (85 molar, 28 premolar teeth) were treated with Spongostan placed in the tooth socket after extraction, spongostan with Chlorhexidine gel and spongostan with tranexamic acid, randomly distributed. After extraction, alveolitis was observed and evaluated prospectively using spongostan, chlorhexidine gel and tranexamic acid in the dental sockets. The researcher checked the participants on the 3rd and 7th days after the tooth extraction. The researcher recorded the pain and edema levels by asking the participants between 0 and 10 using the Visual Analogue Scale (VAS). The researcher filled in the forms for the presence of halitosis, trismus and exposed bone socket on the 3rd and 7th days (YES-NO). Permanent analyzes of the study were created with the SPSS package program.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals between the ages of 18-65
2. Molar and premolar teeth with extraction indication

Exclusion Criteria:

1. Against drugs or substances to be used in surgery (articaine, tranexamic acid, chlorhexidine) have allergies,
2. Those who used antibiotics 30 days before the dental extraction,
3. Clinical and radiological examinations in the operation area 30 days before dental extraction and/or on the day of the procedure.

   Any signs of pathology and infection (such as periapical pathology, pericoronitis),
4. Those who routinely use oral antiseptics,
5. Systemic fever, absence of growth such as lymphadenopathy (LAP),
6. Women are lactating or pregnant,
7. Using oral contraceptives,
8. Procedures that were not attended to control appointments (day 3-7) were not included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-05-26 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
pain | 3.-7. days
  scored on visual analog scale from 0 to 10
edema | 3. day - 7. day
  scored on visual analog scale from 0 to 10
trismus | 3. day - 7. day
  marked yes or no based on clinical examination
halitosis | 3. day - 7. day
  marked yes or no based on clinical examination
alveolar osteitis | 3. day - 7. day
  marked yes or no based on clinical examination
smoking habit | operated day
  marked yes or no based on anamnesis
age | operated day
  marked yes or no based on anamnesis
tooth type | operated day
  marked yes or no based on clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Gümrükçü, Study Director — Recep Tayyip Erdogan University
Locations (1):
- Recep Tayyip Erdoğan University, Rize, Turkey (Türkiye)

REFERENCES:
- [Derived] Gumrukcu Z, Karabag M, Guven SE. The effects of chlorhexidine gel and tranexamic acid application after tooth extraction on the risk of alveolar osteitis formation: a double blind clinical study. Clin Oral Investig. 2024 Aug 21;28(9):494. doi: 10.1007/s00784-024-05886-x. PMID 39167305